CLINICAL TRIAL: NCT03789721
Title: Adrenoleukodystrophy National Registry Study
Status: Recruiting | Type: Observational
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 2019NTLS027; MT2019-01 (Other: University of Minnesota Masonic Cancer Center)
Record Dates: First submitted 2018-12-14; First posted 2018-12-31 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: ALD (Adrenoleukodystrophy); Adrenoleukodystrophy; Cerebral Adrenoleukodystrophy
Keywords: Registry, VLCFA, ABCD1, X-chromosome
MeSH Terms: conditions — Adrenoleukodystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 99 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adrenoleukodystrophy: All patients living in the United States diagnosed with adrenoleukodystrophy, either by newborn screen, based on family history or otherwise, are eligible to participate in this study.
  Interventions: Other: Medical Record Abstraction; Other: Biospecimen Sample Collection

INTERVENTIONS:
Other: Medical Record Abstraction — Collect clinical and epidemiological data through medical record abstraction and self-reported questionnaire survey semi-annually.
Other: Biospecimen Sample Collection — Collect research samples, when feasible for those diagnosed with ALD.

SUMMARY:
The aim of this registry to understand the natural history and disease progression in ALD and potentially develop bio-markers using the biospecimens collected using this registry.

DETAILED DESCRIPTION:
This is a prospective, non-therapeutic protocol designed to create and maintain a registry of participants with Adrenoleukodystrophy (ALD) and known/presumed mutation for ALD. This study also involves maintaining a prospective biorepository to collect and store buccal swab, blood, stool and urine samples as well. In this protocol, pediatric (including infants), adolescents and adult patients with confirmed or presumed ALD (based on positive VLCFA testing and/or confirmed mutation) will be offered potential study participation. Additionally, presumed mutation for ALD (based on pedigree or confirmed mutation) will be offered potential study participation. After appropriate consent (online or in-person), subjects will be requested to provide a medical history (with authorization of release of medical records), longitudinal biospecimens, and permission to perform laboratory analyses on these samples. The overall goal is to understand the natural disease course in affected and unaffected patients (identified patients and relatives with a diagnosis of ALD), as well as women with ALD to assemble a resource of clinical, medical, and biological data from the participants. This study also aims to understand the outcomes of this disease, as well as possibly develop biomarkers to identify prognostic markers for disease progression, which may help develop effective interventions. The biospecimen bank and registry will provide access to samples and data for the ongoing studies as well as will provide an important resource for the future research.

ELIGIBILITY:
Inclusion Criteria

* Age 0 - 100
* ALD patients or family member meeting any of the following criteria:

  * Any patient diagnosed with ALD (confirmed by positive VLCFA testing and/or genetic mutation).
  * Known or presumed mutation with ALD based on pedigree or confirmed mutation in ABCD1 gene
* Participants living in the United States and territories

Exclusion Criteria

* Patients diagnosed with ALD who lack the capacity to consent/assent AND do not have a designated legally authorized representative or guardian.
* Patients who have undergone BMT or other cellular therapy .
* Patients not fluent in English who are unable to consent in-person at the BMT Journey Clinic.
* Patients who are illiterate
* Patient determined by the PI or designee to be unlikely to complete required study components (due to language barriers, compliance issues, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: participants with Adrenoleukodystrophy (ALD) and known/presumed mutation for ALD.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Collect Clinical and Epidemiological Data | 10 Years
  Collect clinical and epidemiological data through medical record abstraction and self-reported questionnaire survey semi-annually.

CONTACTS AND LOCATIONS:
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States